CLINICAL TRIAL: NCT01748474
Title: Effect of Short-term Oxygen Therapy on Cardiopulmonary Exercise Capacity in Patients With Pulmonary Arterial and Chronic Thromboembolic Pulmonary Hypertension
Brief Title: Effect of Short-term Oxygen During CPET in Pulmonary Hypertension
Acronym: ExOx-CPET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: KEK-ZH-NR. 2012-0251
Record Dates: First submitted 2012-10-04; First posted 2012-12-12 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Pulmonary Arterial and Chronic Thromboembolic Pulmonary Hypertension; Chronic Cardiorespiratory Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supplemental oxygen (Experimental): Supplemental oxygen will be applied via a mask during CPET
  Interventions: Procedure: Supplemental oxygen via a mask
- Sham room air (Placebo Comparator): Room air will be applied similarly to oxygen
  Interventions: Procedure: Supplemental oxygen via a mask

INTERVENTIONS:
Procedure: Supplemental oxygen via a mask

SUMMARY:
In a randomized, sham-controlled trial the investigators will test whether supplemental oxygen given during cardiopulmonary exercise testing will improve exercise performance and physiological parameters in patients with pulmonary arterial or chronic thromboembolic pulmonary hypertension.

ELIGIBILITY:
Inclusion criteria:

* diagnosis of pulmonary arterial hypertension class I and IV (according to the latest WHO classification scheme of Dana Point 2008)
* on optimized medical therapy and in stable condition for at least 4 week
* desaturate in the 6 minute walking test by at least 4% to values <92%

Exclusion criteria:

* unstable conditions
* pregnant women
* patients with pulmonary venous hypertension
* patients with relevant concomitant lung disease and severe daytime hypoxemia

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-12; Primary Completion 2016-03 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Watt | 1 day
exercise time | 1 day

SECONDARY OUTCOMES:
Peak oxygen uptake | 1 day
Respiratory exchange ratio | 1 day
ventilatory equivalent of carbon dioxide (VE/VCO2) slope | 1 day
end-tidal pressures of carbon dioxide (PET CO2) | 1 day
Changes in arterial blood parameters | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Ulrich Somaini, MD, Principal Investigator — University Hospital Zurich, Division of Pneumology
Locations (1):
- University Hospital Zurich, Division of Pneumology, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Ulrich S, Hasler ED, Saxer S, Furian M, Muller-Mottet S, Keusch S, Bloch KE. Effect of breathing oxygen-enriched air on exercise performance in patients with precapillary pulmonary hypertension: randomized, sham-controlled cross-over trial. Eur Heart J. 2017 Apr 14;38(15):1159-1168. doi: 10.1093/eurheartj/ehx099. PMID 28329240